CLINICAL TRIAL: NCT01034878
Title: Phase II Study of Sunitinib in Metastatic Renal Cancer With Non-clear Cell Histology
Brief Title: Sunitinib in Metastatic Renal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2008-004
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): 50 mg once daily 6 weeks cycle 4 weeks on and 2 weeks off
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib will be administered orally at a dose of 50 mg once daily, in six weeks cycles consisting of 4 weeks of treatment followed by 2 weeks without treatment.
  Other Names: Sutent

SUMMARY:
Sunitinib is the registered treatment for first-line therapy of metastatic clear-cell carcinoma of the kidney.Data from the Expanded Access Study have shown activity also in non-clear cell renal cancer (NCCRC). The aim of this study is to prospectively evaluate the anti-tumor activity and safety of sunitinib as a first-line therapy in metastatic NCCRC patients.

DETAILED DESCRIPTION:
This is a prospective, open label, multicenter phase II study to evaluate efficacy of Sunitinib (in advanced/metastatic renal cancer with non-clear cell histology (papillary or chromophobe).

Sunitinib will be administered orally at a dose of 50 mg once daily, in six weeks cycles consisting of 4 weeks on treatment followed by 2 weeks off.

Treatment with the study drug will continue until tumor progression or unacceptable toxicity.

The planned total sample size for this study is 55 patients. Approximately 10 study sites will be involved.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of metastatic renal cancer with non-clear cell
* No previous treatment

Exclusion Criteria:

* Prior treatment with an antiangiogenetic compound
* Symptomatic and/or unstable pre-existing brain metastases
* Severe or uncontrolled cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The antitumor activity in terms of progression free survival | two years

SECONDARY OUTCOMES:
To evaluate the objective response rate | two years
To evaluate the toxicity and the safety profile | two years
To evaluate the overall survival | two years

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinco Humanitas, Rozzano, Milano, Italy